CLINICAL TRIAL: NCT04075448
Title: The Acute Effect of a Walnut Intervention on Cognitive Performance , Brain Activation, and Serum Markers of Inflammation in Young Adults
Brief Title: The Acute Effect of a Walnut Intervention on Cognitive Performance, Brain Activation, and Serum Markers of Inflammation in Young Adults
Acronym: WalCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: California Walnut Commission (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Chair of Neuroscience, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RDG-005
Record Dates: First submitted 2019-08-07; First posted 2019-08-30 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cognitive Change; Mood; Inflammatory Response; Brain Derived Neurotrophic Factor Level; Satiety
Keywords: Flavonoid; Omega 3 Fatty Acid

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to both the walnut and control conditions in a randomised order.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be aware the possible contents of each treatment, however, neither the participants or investigators will be aware of which treatment the participants are receiving at the point of testing. All analysis will be performed in relation to a treatment code which will only be revealed once analysis is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - 50g Walnut (Experimental): Control condition followed by experimental condition.
  Interventions: Other: Control; Other: 50 g Walnut
- 50 g Walnut - Control (Experimental): Experimental condition followed by control condition.
  Interventions: Other: Control; Other: 50 g Walnut

INTERVENTIONS:
Other: Control — 100 grams breakfast cereal
Other: 50 g Walnut — 50 grams walnuts mixed with 50 gram breakfast cereal.

SUMMARY:
This study investigates the effect of acute walnut consumption on the cognitive behaviour, mood, brain activation, and markers of inflammation in young adults. In a within subjects design participants will receive a 50 g walnut or placebo intervention in a randomised order with a one week washout between interventions.

DETAILED DESCRIPTION:
Participants will attend two test session days separated by a 7 day wash out period. The procedure on each day will be identical save for the intervention breakfast which will either be a walnut rich muesli containing 50g walnut and 50g mixed cereal ingredients (active intervention), or control muesli containing 100g mixed cereal ingredients (placebo intervention). The order of intervention will be randomised such that 50% of participants receive the active intervention during visit 1 and 50% during visit 2. Participants will be required to follow a low flavonoid diet for 48 hours in advance of testing and to fast (water only) for the final 12 hours of this period. The test day will be 8hrs in total starting at 0830.

Cognitive Measures: There will be four cognitive task battery sessions taking place at baseline, then 2, 4, and 6 hours following intervention. The cognitive battery will last for 30 minutes and include:

* Auditory Verbal Learning Task (AVLT) - Participants hear and recall a list of 15 words on 8 occasions followed by a forced choice visual recognition task (10 minutes duration).
* Modified Attention Network Task (MANT) - Participants view different arrays of arrows displayed on a monitor and respond by indicating the direction of the arrow closest to a central fixation point (8 minutes duration).
* Switching Task - Participants view eight equally spaced radii of circle displayed in such a way that there are four equally spaced segments above and below a bold line. Stimulus digits selected from between 1 - 9 (excluding 5) appear in each segment in turn. Participants respond to digits above the bold line in terms of whether they are odd or even and below the bold line in terms of whether they are above or below the number 5 (10 minutes duration).
* PANAS-NOW - This measure of trait mood will be completed at the beginning and end of each task battery giving a total of 8 measurements across the day. Participants rate the extent to which they are experiencing 20 different emotions on a 5-point Likert scale ranging from 'very slightly' to 'very much' (1 minute duration).

EEG: All participants will be tested in our dedicated lab within the Reading University Centre for Integrative Neuroscience and Neurodynamics using the Brain Products EEG system with 32 channel active electrode caps. At Baseline, 2, 4 and 6 hrs waveband PSD data will be recorded during all tasks with specific attention being paid to the theta bandwidth during the AVLT and gamma bandwidth during the executive function tasks. ERP data, anchored to each trial of the executive function tasks, will also be considered with specific attention being given to latency and strength of N1 and P3 peaks.

Bloods: Participants will have bloods taken twice on each test visit with a draw being taken from each arm. The initial draw will be taken immediately prior to the baseline task battery and then immediately prior to either the 2, 4 or 6 hr session with the second draw time being randomised in such a way that 16 participants will have blood drawn at 2hrs, 16 at 4hrs, and 16 at 6hrs. Following each draw, the blood samples will be left to clot for 30-60 minutes. The serum will be separated via centrifuge and stored at at -80°C until analysis is complete. Whole blood samples will not be stored at any point during the study. Blood serum will be analysed for anti-inflammatory ability, as well as levels of BDNF, a signalling protein known to be positively related to memory function. To determine possible mechanisms of action of walnut components through which the walnut polyphenols produce their beneficial effects, microglial cells from rats will be exposed to serum from participants in both walnut and placebo conditions prior to exposure to an inflammatory challenge (LPS). Markers of inflammation will then be assessed including extracellular release of nitric oxide (NO) and tumor necrosis factor-alpha (TNF-α) as well as intracellular levels of inducible nitrous oxide synthase (iNOS) and cyclooxygenase-2 (COX-2). We will then determine if those subjects with the most protective serum in the cell model are those with the better cognitive performance.

Appetite Measures: Ratings of subjective appetite and fullness will be taken using visual analogue scales after baseline, breakfast, and each of the remaining test sessions. As a further measure of satiety, weighted food measurements will be taken before and after consumption of the standard low flavonoid/PUFA lunch (given immediately after task battery session 3 at 1330) to ascertain total food consumption.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal or corrected hearing and vision

Exclusion Criteria:

* Smoker.
* Allergic to treatment contents.
* Currently on medication which may interfere with the treatment
* Anaemic

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Delayed Recall | 2 hours following intervention.
  AVLT - Recall of a previously presented list of words following a 25 minute delay.
Delayed Recall | 4 hours following intervention.
  AVLT - Recall of a previously presented list of words following a 25 minute delay.
Delayed Recall | 6 hours following intervention.
  AVLT - Recall of a previously presented list of words following a 25 minute delay.
Word Recognition | 2 hours following intervention.
  AVLT - Visual Recognition of a previously presented list of words following a 25 minute delay.
Word Recognition | 4 hours following intervention.
  AVLT - Visual Recognition of a previously presented list of words following a 25 minute delay.
Word Recognition | 6 hours following intervention.
  AVLT - Visual Recognition of a previously presented list of words following a 25 minute delay.
Response interference accuracy | 2 hours following intervention.
  Accuracy performance on the Modified Attention Network Task
Response interference accuracy | 4 hours following intervention.
  Accuracy performance on the Modified Attention Network Task
Response interference accuracy | 6 hours following intervention.
  Accuracy performance on the Modified Attention Network Task
Response interference reaction time | 2 hours following intervention
  Reaction time performance on the Modified Attention Network Task
Response interference reaction time | 4 hours following intervention
  Reaction time performance on the Modified Attention Network Task
Response interference reaction time | 6 hours following intervention
  Reaction time performance on the Modified Attention Network Task
Switching Task Accuracy | 2 hours following intervention
  Accuracy performance on the switching task
Switching Task Accuracy | 4 hours following intervention
  Accuracy performance on the switching task
Switching Task Accuracy | 6 hours following intervention
  Accuracy performance on the switching task
Switching Task reaction time | 2 hours following intervention
  Reaction time performance on the switching task
Switching Task reaction time | 4 hours following intervention
  Reaction time performance on the switching task
Switching Task reaction time | 6 hours following intervention
  Reaction time performance on the switching task
N2 | 2 hours following intervention
  Change in ERP measure of N2 latency and amplitude
N2 | 4 hours following intervention
  Change in ERP measure of N2 latency and amplitude
N2 | 6 hours following intervention
  Change in ERP measure of N2 latency and amplitude
P3 | 2 hours following intervention
  Change in ERP measure of P3 latency and amplitude
P3 | 4 hours following intervention
  Change in ERP measure of P3 latency and amplitude
P3 | 6 hours following intervention
  Change in ERP measure of P3 latency and amplitude
Inflammatory Measure of nitrous oxide, tumor necorsis factor-alpha, inducible nitrous oxide synthase, and tumor necrosis facor-alpha. | 2 hours following intervention
  Change in blood serum markers of inflammation
Inflammatory Measure of nitrous oxide, tumor necorsis factor-alpha, inducible nitrous oxide synthase, and tumor necrosis facor-alpha. | 4 hours following intervention
  Change in blood serum markers of inflammation
Inflammatory Measure of nitrous oxide, tumor necorsis factor-alpha, inducible nitrous oxide synthase, and tumor necrosis facor-alpha. | 6 hours following intervention
  Change in blood serum markers of inflammation
BDNF | 2 hours following intervention
  Change in blood serum levels of BDNF
BDNF | 4 hours following intervention
  Change in blood serum levels of BDNF
BDNF | 6 hours following intervention
  Change in blood serum levels of BDNF

SECONDARY OUTCOMES:
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption (Flint et al., 2000). | 2 hours following intervention.
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger - taken as a positive outcome, less satiety - taken as a negative outcome, less fullness - taken as a negative outcome, and less desire for prospective food consumption - taken as a positive.
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption (Flint et al., 2000). | 4 hours following intervention.
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger - taken as a positive outcome, less satiety - taken as a negative outcome, less fullness - taken as a negative outcome, and less desire for prospective food consumption - taken as a positive.
Visual analogue measure of hunger, satiety, fullness, and prospective food consumption (Flint et al., 2000). | 6 hours following intervention.
  Satiety Measure recorded on a 100 millimetre scale. Scores closer to 0 millimetres indicate less hunger - taken as a positive outcome, less satiety - taken as a negative outcome, less fullness - taken as a negative outcome, and less desire for prospective food consumption - taken as a positive.
EEG Spectral Analysis. | 2 hours following intervention.
  Changes in Power for Alpha, Beta, Gamma, Delta, and Theta bands during performance of each cognitive task.
EEG Spectral Analysis. | 4 hours following intervention.
  Changes in Power for Alpha, Beta, Gamma, Delta, and Theta bands during performance of each cognitive task.
EEG Spectral Analysis. | 6 hours following intervention.
  Changes in Power for Alpha, Beta, Gamma, Delta, and Theta bands during performance of each cognitive task.
Immediate Recall | 2 hours following intervention
  AVLT - Immediate recall following first presentation of the word list
Immediate Recall | 4 hours following intervention
  AVLT - Immediate recall following first presentation of the word list
Immediate Recall | 6 hours following intervention
  AVLT - Immediate recall following first presentation of the word list
Word Learning | 2 hours following intervention
  AVLT - Area under the curve for first five word list recalls.
Word Learning | 4 hours following intervention
  AVLT - Area under the curve for first five word list recalls.
Word Learning | 6 hours following intervention
  AVLT - Area under the curve for first five word list recalls.
Total Recall | 2 hours following intervention.
  AVLT - Sum of first 5 word list recalls.
Total Recall | 4 hours following intervention.
  AVLT - Sum of first 5 word list recalls.
Total Recall | 6 hours following intervention.
  AVLT - Sum of first 5 word list recalls.
Final Acquisition | 2 hours following intervention
  AVLT - Immediate recall following final presentation of the word list
Final Acquisition | 4 hours following intervention
  AVLT - Immediate recall following final presentation of the word list
Final Acquisition | 6 hours following intervention
  AVLT - Immediate recall following final presentation of the word list
Interference List Recall | 2 hours following intervention.
  AVLT - Immediate recall of second (interference) list.
Interference List Recall | 4 hours following intervention.
  AVLT - Immediate recall of second (interference) list.
Interference List Recall | 6 hours following intervention.
  AVLT - Immediate recall of second (interference) list.

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Williams, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full dataset will be anonymized and made available on the University of Reading Research Data Archive.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be become available upon publication of study findings. Once published, the data will remain permanently available.
Access Criteria: The data will be Open Access and licensed as Creative Commons: Attribution 4.0

REFERENCES:
- [Background] Bell L, Lamport DJ, Butler LT, Williams CM. A Review of the Cognitive Effects Observed in Humans Following Acute Supplementation with Flavonoids, and Their Associated Mechanisms of Action. Nutrients. 2015 Dec 9;7(12):10290-306. doi: 10.3390/nu7125538. PMID 26690214
- [Background] Carey AN, Fisher DR, Joseph JA, Shukitt-Hale B. The ability of walnut extract and fatty acids to protect against the deleterious effects of oxidative stress and inflammation in hippocampal cells. Nutr Neurosci. 2013 Jan;16(1):13-20. doi: 10.1179/1476830512Y.0000000023. Epub 2012 Dec 4. PMID 23321679
- [Background] Fisher DR, Poulose SM, Bielinski DF, Shukitt-Hale B. Serum metabolites from walnut-fed aged rats attenuate stress-induced neurotoxicity in BV-2 microglial cells. Nutr Neurosci. 2017 Feb;20(2):103-109. doi: 10.1179/1476830514Y.0000000150. Epub 2016 Mar 2. PMID 25153536
- [Background] Gomez-Pinilla F. Brain foods: the effects of nutrients on brain function. Nat Rev Neurosci. 2008 Jul;9(7):568-78. doi: 10.1038/nrn2421. PMID 18568016
- [Background] Haider S, Batool Z, Tabassum S, Perveen T, Saleem S, Naqvi F, Javed H, Haleem DJ. Effects of walnuts (Juglans regia) on learning and memory functions. Plant Foods Hum Nutr. 2011 Nov;66(4):335-40. doi: 10.1007/s11130-011-0260-2. PMID 22048906
- [Background] Martinez-Lapiscina EH, Clavero P, Toledo E, Estruch R, Salas-Salvado J, San Julian B, Sanchez-Tainta A, Ros E, Valls-Pedret C, Martinez-Gonzalez MA. Mediterranean diet improves cognition: the PREDIMED-NAVARRA randomised trial. J Neurol Neurosurg Psychiatry. 2013 Dec;84(12):1318-25. doi: 10.1136/jnnp-2012-304792. Epub 2013 May 13. PMID 23670794
- [Background] Miller MG, Thangthaeng N, Poulose SM, Shukitt-Hale B. Role of fruits, nuts, and vegetables in maintaining cognitive health. Exp Gerontol. 2017 Aug;94:24-28. doi: 10.1016/j.exger.2016.12.014. Epub 2016 Dec 21. PMID 28011241
- [Background] Nooyens AC, Bueno-de-Mesquita HB, van Boxtel MP, van Gelder BM, Verhagen H, Verschuren WM. Fruit and vegetable intake and cognitive decline in middle-aged men and women: the Doetinchem Cohort Study. Br J Nutr. 2011 Sep;106(5):752-61. doi: 10.1017/S0007114511001024. Epub 2011 Apr 11. PMID 21477405
- [Background] O'Brien J, Okereke O, Devore E, Rosner B, Breteler M, Grodstein F. Long-term intake of nuts in relation to cognitive function in older women. J Nutr Health Aging. 2014 May;18(5):496-502. doi: 10.1007/s12603-014-0014-6. PMID 24886736
- [Background] Perez-Cano FJ, Castell M. Flavonoids, Inflammation and Immune System. Nutrients. 2016 Oct 21;8(10):659. doi: 10.3390/nu8100659. PMID 27775647
- [Background] Poulose SM, Bielinski DF, Shukitt-Hale B. Walnut diet reduces accumulation of polyubiquitinated proteins and inflammation in the brain of aged rats. J Nutr Biochem. 2013 May;24(5):912-9. doi: 10.1016/j.jnutbio.2012.06.009. Epub 2012 Aug 20. PMID 22917841
- [Background] Pribis P, Bailey RN, Russell AA, Kilsby MA, Hernandez M, Craig WJ, Grajales T, Shavlik DJ, Sabate J. Effects of walnut consumption on cognitive performance in young adults. Br J Nutr. 2012 May;107(9):1393-401. doi: 10.1017/S0007114511004302. Epub 2011 Sep 19. PMID 21923981
- [Background] Ros E, Hu FB. Consumption of plant seeds and cardiovascular health: epidemiological and clinical trial evidence. Circulation. 2013 Jul 30;128(5):553-65. doi: 10.1161/CIRCULATIONAHA.112.001119. No abstract available. PMID 23897849
- [Background] Sanchez-Villegas A, Galbete C, Martinez-Gonzalez MA, Martinez JA, Razquin C, Salas-Salvado J, Estruch R, Buil-Cosiales P, Marti A. The effect of the Mediterranean diet on plasma brain-derived neurotrophic factor (BDNF) levels: the PREDIMED-NAVARRA randomized trial. Nutr Neurosci. 2011 Sep;14(5):195-201. doi: 10.1179/1476830511Y.0000000011. PMID 22005283
- [Background] Valls-Pedret C, Sala-Vila A, Serra-Mir M, Corella D, de la Torre R, Martinez-Gonzalez MA, Martinez-Lapiscina EH, Fito M, Perez-Heras A, Salas-Salvado J, Estruch R, Ros E. Mediterranean Diet and Age-Related Cognitive Decline: A Randomized Clinical Trial. JAMA Intern Med. 2015 Jul;175(7):1094-1103. doi: 10.1001/jamainternmed.2015.1668. PMID 25961184
- [Background] Willis LM, Shukitt-Hale B, Cheng V, Joseph JA. Dose-dependent effects of walnuts on motor and cognitive function in aged rats. Br J Nutr. 2009 Apr;101(8):1140-4. doi: 10.1017/S0007114508059369. PMID 18778529
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749